CLINICAL TRIAL: NCT02633228
Title: Evaluation of the Visual Acuity After the Implantation of an Oculentis +2.0 Diopters (Torical) Bifocal Intraocular Lens (MplusX (Toric) LU-313 MF20T/LS-313 MF20) in the Distance Dominant Eye, in Combination With a +3.0 Diopters Oculentis Bifocal Intraocular Lens (MplusX (Toric) LU-313 MF30T/LS-313 MF30) in the Fellow Eye.
Brief Title: Visual Acuity After the Combined Binocular Implantation of +2.0 Diopters and +3.0 Diopters Oculentis Multifocal Intraocular Lenses.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PD Dr. med. Eckart Bertelmann (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Eckart Bertelmann, Senior Consultant, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA2/129/14
Record Dates: First submitted 2015-12-14; First posted 2015-12-17 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Cataract
Keywords: Multifocal Intraocular Lens; Binocular Trifocality; Cataract Surgery; Spectacle Independence; Intermediate Vision; Photopic Vision; Mesopic Vision; Scotopic Vision; Binocular Vision
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Binocular cataract surgery with phacoemulsification and implantation of multifocal intraocular lenses — Binocular implantation of the combination of Oculentis® MplusX® multifocal intraocular lenses with an addition of +2.0 D in the distance-dominant eye and +3.0 D in the fellow eye.
  Other Names: Oculentis® MplusX® multifocal intraocular lenses with an addition of +2.0 D (LU-313 MF20T/LS-313 MF20) and +3.0 D (LU-313 MF30T/LS-313 MF30) are used.

SUMMARY:
The objective of this study is to assess the visual outcome after the combined binocular implantation of +2.0 D and +3.0 D refractive multifocal intraocular lenses.

DETAILED DESCRIPTION:
Bifocal multifocal intraocular lenses (MIOL) are effective in achieving good uncorrected visual acuities in the distance and the near. However, the intermediate vision is of increasing relevance for everyday's life. Several multifocal intraocular lenses have been developed to improvement intermediate vision. Nonetheless, those systems still possess adverse photic effects and do not garantuee spectacle independence. Therefore, the combination of a lower-addition bifocal intraocular lense in the distance-dominant eye with a higher-addition bifocal intraocular lense in the fellow-eye might be a promising approach to address these drawbacks of current binocular and trifocal intraocular lenses.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant cataract
* endothelial cell count: patients aged 18-75 years: > 1000 cells/mm2; patients > 75 years: > 750 cells/mm2
* absence of vision-limiting corneal or retinal comorbidities
* capability to understand the informed consent

Exclusion Criteria:

* expected postoperative astigmatism > 0.75 diopters
* irregular astigmatism
* dilated pupil diameter < 3 mm
* corneal and fundus abnormalities that might cause visual impairments
* inability to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Visual acuities in the far, intermediate and near | 1 month
  Visual acuities are tested under photopic conditions at 5 m, intermediate (80 cm) and patient-preferred near distance (≈ 40 cm).
Visual acuities in the far, intermediate and near | 3 months
  Visual acuities are tested under photopic conditions at 5 m, intermediate (80 cm) and patient-preferred near distance (≈ 40 cm).
Mesopic vision | 1 month
  Mesopic visual acuities are tested under high-contrast, low-contrast and low-contrast with glare.
Mesopic vision | 3 months
  Mesopic visual acuities are tested under high-contrast, low-contrast and low-contrast with glare.
Scotopic contrast sensitivity | 1 month
  Scotopic contrast sensitivity are tested at 0.1 cd/m2, 0.032 cd/m2 and 0.1 cd/m2 with glare.
Scotopic contrast sensitivity | 3 months
  Scotopic contrast sensitivity are tested at 0.1 cd/m2, 0.032 cd/m2 and 0.1 cd/m2 with glare.

SECONDARY OUTCOMES:
Spectacle independence in the far, intermediate and near | 3 months
  Spectacle independence as stated by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Eckart Bertelmann, MD, PhD, Principal Investigator — Charité - University Medicine Berlin, Department of Ophthalmology
Locations (1):
- Charité - University Medicine Berlin, Department of Ophthalmology, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alio JL, Plaza-Puche AB, Javaloy J, Ayala MJ, Vega-Estrada A. Clinical and optical intraocular performance of rotationally asymmetric multifocal IOL plate-haptic design versus C-loop haptic design. J Refract Surg. 2013 Apr;29(4):252-9. doi: 10.3928/1081597X-20130318-04. PMID 23557223
- [Background] Bonaque-Gonzalez S, Rios S, Amigo A, Lopez-Gil N. Influence on Visual Quality of Intraoperative Orientation of Asymmetric Intraocular Lenses. J Refract Surg. 2015 Oct;31(10):651-7. doi: 10.3928/1081597X-20150922-01. PMID 26469073
- [Background] Garcia-Domene MC, Felipe A, Peris-Martinez C, Navea A, Artigas JM, Pons AM. Image quality comparison of two multifocal IOLs: influence of the pupil. J Refract Surg. 2015 Apr;31(4):230-5. doi: 10.3928/1081597X-20150319-02. PMID 25884577
- [Background] Alio JL, Plaza-Puche AB, Pinero DP. Rotationally asymmetric multifocal IOL implantation with and without capsular tension ring: refractive and visual outcomes and intraocular optical performance. J Refract Surg. 2012 Apr;28(4):253-8. doi: 10.3928/1081597X-20120314-01. PMID 22496436
- [Background] Munoz G, Albarran-Diego C, Javaloy J, Sakla HF, Cervino A. Combining zonal refractive and diffractive aspheric multifocal intraocular lenses. J Refract Surg. 2012 Mar;28(3):174-81. doi: 10.3928/1081597X-20120215-02. PMID 22373031